CLINICAL TRIAL: NCT03278808
Title: A Phase 2a Open Label Study of the Safety and Efficacy of a Single Dose of Weekly Chloroquine (CQ) and Azithromycin (AZ) Administered in Combination for Malaria Prophylaxis in Healthy Adults Challenged With 7G8 Chloroquine-Resistant Plasmodium Falciparum in a Controlled Human Malaria Infection (CHMI) Model
Brief Title: Chloroquine (CQ) and Azithromycin (AZ) Combination for Malaria Prophylaxis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The IND has been withdrawn from FDA
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-16-06
Record Dates: First submitted 2017-08-24; First posted 2017-09-12 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Chloroquine; atovaquone, proguanil drug combination

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to either the CQ/AZ group (Group 1 of 15 subjects: 2 g AZ (Zithromax) plus 300 mg CQ base weekly for 6 weeks), or the CQ control group (Group 2 of 8 subjects: 300 mg chloroquine base weekly for 6 weeks)
Masking Description: Because placebo for both products is difficult to obtain and because the primary endpoint of symptomatic parasitemia is an objective measure, treatment will be open-label. Microscopists reading the smears will be blinded to the group, but will be aware of whether or not a particular sample is from a symptomatic subject.
  Although symptoms are a subjective measure and part of the primary endpoint of symptomatic parasitemia, subjects will not be told if they are parasitemic prior to treatment initiation thus making symptomatic complaints and this endpoint more reliable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Chloroquine-Azithromycin (CQ/AZ ) Group (Experimental): Subjects will receive experimental intervention of 300mg of CQ orally (PO) and 2g of AZ PO weekly for 6 weeks
  Interventions: Drug: Chloroquine-Azithromycin (CQ/AZ)
- Chloroquine (CQ) Group (Active Comparator): Subjects will only receive 300mg of CQ orally (PO) weekly for 6 weeks
  Interventions: Drug: Chloroquine (CQ)
- CHMI Group - atovaquone-proguanil (Malarone®) (Other): All subjects will participate in the Controlled Human Malaria Infection (CHMI) and will be required to stay at a hotel for evaluation for a maximum of 14 nights starting 7 days after the challenge. A standard dose of atovaquone-proguanil (Malarone®) will be administered to all symptomatic parasitemic subjects under directly observed treatment.
  Interventions: Drug: atovaquone-proguanil (Malarone®)

INTERVENTIONS:
Drug: Chloroquine-Azithromycin (CQ/AZ) — Chloroquine-Azithromycin (CQ/AZ); Chloroquine (CQ) 300mg and 2g of azithromycin (AZ) given orally
  Other Names: CQ/AZ
  Arms: Chloroquine-Azithromycin (CQ/AZ ) Group
Drug: Chloroquine (CQ) — Chloroquine (CQ); 300 mg of CQ only given orally
  Other Names: CQ
  Arms: Chloroquine (CQ) Group
Drug: atovaquone-proguanil (Malarone®) — All subjects will participate in the Controlled Human Malaria Infection (CHMI) and will be required to stay at a hotel for evaluation for a maximum of 14 nights starting 7 days after the challenge. A standard dose of atovaquone-proguanil (Malarone®) will be administered to all symptomatic parasitemic subjects under directly observed treatment.
  Arms: CHMI Group - atovaquone-proguanil (Malarone®)

SUMMARY:
This is an open label, Phase 2 study with controlled human malaria infection (CHMI). Twenty three subjects will be enrolled into 2 groups (15 subjects in the Chloroquine-Azithromycin [CQ/AZ] Intervention Group, and 8 subjects in the Chloroquine [CQ] Group). The CQ/AZ Group will receive experimental intervention of 300 mg of CQ and 2 g of azithromycin (AZ). The CQ Group will receive 300 mg of CQ only. All subjects will participate in the CHMI and will be required to stay at a hotel for evaluation for a maximum of 14 nights starting 7 days after the challenge. A standard dose of atovaquone-proguanil (Malarone®) will be administered to all symptomatic parasitemic subjects under directly observed treatment.

DETAILED DESCRIPTION:
This study is a Phase 2, open-label study of the combination of a single dose-level of AZ (Zithromax) plus CQ given weekly as a prophylaxis against CQ-resistant P falciparum in healthy adults. After signing informed consent, subjects will undergo screening procedures between Day -77 to Day -18. If enrolled, subjects who are still eligible at Study Day -18 will be randomized to either the CQ/AZ group (Group 1 of 15 subjects: 2 g AZ (Zithromax) plus 300 mg CQ base weekly for 6 weeks), or the CQ control group (Group 2 of 8 subjects: 300 mg chloroquine base weekly for 6 weeks) and start intervention on Study Day -17. The rationale for the CQ control group to receive CQ is to show that the strain utilized (7G8) is indeed chloroquine resistant in humans: we expect all of the subjects in the CQ control group to become symptomatically parasitemic. If 3 or more subjects in the CQ control group do not become symptomatic with malaria, the CHMI will be considered uncontrolled either due to 7G8 not being CQ-resistant, or the parasite not being infective.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (male or non-pregnant, non-lactating female) 18 to 50 years of age (inclusive) at the time of screening.
* If the subject is female:

  1. Non-childbearing potential (ie., either surgically sterilized (bilateral tubal ligation, tubes tied, hysterectomy, removal of the uterus, bilateral oophorectomy, removal of both ovaries) at least 6 months before dosing) or one year post menopausal), abstinent or using adequate contraceptive precautions (eg, intrauterine contraceptive device; oral contraceptives; diaphragm, cervical cap, or condom in combination with contraceptive jelly, cream or foam; Norplant® or Depo-Provera®) from 3 months prior to this study through 56 days after challenge
  2. A negative pregnancy test at the time of enrollment
* Free of significant health problems as established by medical history, laboratory, and clinical examination before entering the study
* Subjects must have low cardiac risk factors according to the NHANES I criteria, medical history and family history, blood pressure measurements, and a normal or normal variant ECG including QTcF no greater than 450 msec for males and 470 msec for females.
* Available to participate in all planned study visits and reachable by phone for duration of study (approximately 4 months).
* Willing to comply with all protocol procedures and time commitments
* No plans to participate in another clinical research study for the duration of this study.
* Written informed consent must be obtained from the subject before screening procedures are performed
* If a subject is active duty military, he or she must obtain approval from his or her supervisor per Walter Reed Army Institute of Research (WRAIR) Policy 11-45
* Subjects must score at least 80% correct on a multiple-choice quiz that assesses their understanding of this study

  1. If they do not score 80% on the initial quiz, the protocol information will be reviewed with them, and they will have the opportunity to retest
  2. If a subject fails to correctly answer 80% of the questions after 2 attempts, he or she will be excluded from the study

Exclusion Criteria:

* Subjects with a history or presence of gastrointestinal, hepatic or renal disease, or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Subjects with a history of retinopathy, sickle cell disease or trait, psoriasis, or porphyria.
* Subjects who take certain prescribed or over the counter (OTC) concomitant medication including: ampicillin, antacids (including kaolin), cimetidine, digoxin, ergot alkaloids, statins (HMG-CoA reductase inhibitors), cyclosporine, warfarin, fluconazole, nelfinavir, or rifabutin, within 2 weeks of dosing start, and during the duration of the study.
* Are known or suspected of drinking too much alcohol (for men, more than 28 standard alcohol drinks and for women more than 21 standard alcohol drinks per week (standard drink is defined as a 12 oz beer, 5 oz glass of wine, or 1.5 oz of distilled spirit)
* Positive urine drug screen for amphetamine, methamphetamine, cocaine, and opioids at screening.
* Subjects who have donated more than 1500 mL (males) or 1000 mL (females) blood in the previous 12 months, including the maximum volume of blood (328 mL) to be taken in this study.
* Subjects who are currently enrolled in another study involving an investigational product, or if recently involved in another clinical trial which has ended, have not received any investigational products within the past 3 months or 5 half-lives (whichever is longer) from the time of screening.
* Any history of malaria infection in the past 3 years.
* History of travel to malaria endemic areas in the 3 months prior to day of challenge, or plans to travel to malaria endemic areas during the duration of the study (56 days post challenge).
* Any history of receiving a malaria vaccine
* History of receipt of malaria prophylaxis during the 2 months prior to day of challenge
* History of use of any antibiotics with significant antimalarial activity (examples include tetracycline, doxycycline, clindamycin, azithromycin, and sulfa drugs) during the course of the study period
* Pregnant (positive β-human chorionic gonadotropin test, β-HCG) or lactating female at screening or plans to become pregnant or breastfeed from the time of enrollment until three months after challenge
* Allergy to antimalarial drugs or use of medications known to interact with CQ
* Significant (e.g., systemic) hypersensitivity reactions to mosquito bites (local hypersensitivity reactions at the site of mosquito bites are not an exclusion criterion)
* History of splenectomy
* Any confirmed or suspected immunodeficiency, including HIV infection, or taking immunosuppressive medications
* Acute or chronic, ally significant, pulmonary, cardiovascular, endocrine, hepatic, or renal functional abnormality, as determined by history, physical examination, or laboratory evaluation
* Chronic or active neurologic disease including seizure disorder and chronic migraine headaches
* Any abnormal baseline laboratory screening tests listed below

  1. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) above twice the upper limit of normal for the reference lab
  2. Creatinine above normal range
  3. Hemoglobin out of normal range
  4. Platelet count out of normal range
  5. Total white blood cell (WBC) count out of normal range Note: If screening lab values are out of the normal range but are expected to be temporary (e.g. due to dehydration), they may be re-assessed one time at the discretion of the investigator.
* Seropositive for Human immunodeficiency virus (HIV) or Hepatitis C virus (HCV) or hepatitis B surface antigen (HBsAg) positive
* An abnormal baseline screening ECG suggestive of cardiac disease as determined by a clinical investigator. QTcF of >450 msec for males and >470 msec for females.
* Any other significant finding that in the opinion of the PI would increase the risk of having an adverse outcome from participating in this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Efficacy: Proportion of subjects free from symptomatic parasitemic subjects | Days 1 thru 56
  CQ/AZ Group will be compared to endpoint in CQ Group by Fisher's Exact Test. Symptomatic is defined as any one of the following solicited adverse events that first occurred concurrent with parasitemia: fever (temperature > 100.4 °F), chills, headache, arthralgia, myalgia, nausea, vomiting, or abdominal pain. Subjects will only undergo malaria treatment after both criteria are met.

SECONDARY OUTCOMES:
Safety: Solicited and unsolicited Adverse Events in each group | Days 1 thru 56
  Groups will be analyzed by descriptive statistics and safety monitoring will be conducted throughout the study
Electrocardiogram baseline vs peak concentration for AZ | Day 11 post challenge, 6 hours after dosing
  QTcF will be analyzed for CQ/AZ Group subjects at presumed field-effective time point (Day 11 post challenge) 6 hours after dosing, which will coincide with time to peak concentration for AZ. This will be compared to baseline reading
Pharmacokinetics: Cmax - comparison for CQ/AZ-Group subjects | Days 11 thru 15
  Cmax will be compared for CQ/AZ-Group subjects who become symptomatic and parasitemic to CQ/AZ-Group subjects who do not become parasitemic.
Pharmacokinetics: Tmax - comparison for CQ/AZ-Group | Days 11 thru 15
  Tmax will be compared for CQ/AZ-Group subjects who become symptomatic and parasitemic to CQ/AZ-Group subjects who do not become parasitemic.
Pharmacokentics: T½ - comparison for CQ/AZ Group | Days 11 thru 15
  T½ will be compared for CQ/AZ-Group subjects who become symptomatic and parasitemic to CQ/AZ-Group
Pharmacokentics: AUC - comparison for CQ/AZ Group | Days 11 thru 15
  Area under the curve (AUC) will be compared for CQ/AZ-Group subjects who become symptomatic and parasitemic to CQ/AZ-Group subjects who do not become parasitemic.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Livezey, MD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (2):
- United States (2):
  - Clinical Research Unit, Uniformed Services University of Health Sciences, Bethesda, Maryland
  - WRAIR, Silver Spring, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heppner DG Jr, Walsh DS, Uthaimongkol N, Tang DB, Tulyayon S, Permpanich B, Wimonwattrawatee T, Chuanak N, Laoboonchai A, Sookto P, Brewer TG, McDaniel P, Eamsila C, Yongvanitchit K, Uhl K, Kyle DE, Keep LW, Miller RE, Wongsrichanalai C. Randomized, controlled, double-blind trial of daily oral azithromycin in adults for the prophylaxis of Plasmodium vivax malaria in Western Thailand. Am J Trop Med Hyg. 2005 Nov;73(5):842-9. PMID 16282291
- [Background] Pereira MR, Henrich PP, Sidhu AB, Johnson D, Hardink J, Van Deusen J, Lin J, Gore K, O'Brien C, Wele M, Djimde A, Chandra R, Fidock DA. In vivo and in vitro antimalarial properties of azithromycin-chloroquine combinations that include the resistance reversal agent amlodipine. Antimicrob Agents Chemother. 2011 Jul;55(7):3115-24. doi: 10.1128/AAC.01566-10. Epub 2011 Apr 4. PMID 21464242
- [Background] Taylor WR, Richie TL, Fryauff DJ, Picarima H, Ohrt C, Tang D, Braitman D, Murphy GS, Widjaja H, Tjitra E, Ganjar A, Jones TR, Basri H, Berman J. Malaria prophylaxis using azithromycin: a double-blind, placebo-controlled trial in Irian Jaya, Indonesia. Clin Infect Dis. 1999 Jan;28(1):74-81. doi: 10.1086/515071. PMID 10028075
- [Background] Yeo AE, Rieckmann KH. Increased antimalarial activity of azithromycin during prolonged exposure of Plasmodium falciparum in vitro. Int J Parasitol. 1995 Apr;25(4):531-2. doi: 10.1016/0020-7519(94)00119-9. PMID 7635629
- [Result] Andersen SL, Oloo AJ, Gordon DM, Ragama OB, Aleman GM, Berman JD, Tang DB, Dunne MW, Shanks GD. Successful double-blinded, randomized, placebo-controlled field trial of azithromycin and doxycycline as prophylaxis for malaria in western Kenya. Clin Infect Dis. 1998 Jan;26(1):146-50. doi: 10.1086/516281. PMID 9455524
- [Result] Biswas S. In-vitro antimalarial activity of azithromycin against chloroquine sensitive and chloroquine resistant Plasmodium falciparum. J Postgrad Med. 2001 Oct-Dec;47(4):240-3. PMID 11832638
- [Result] Dunne MW, Singh N, Shukla M, Valecha N, Bhattacharyya PC, Dev V, Patel K, Mohapatra MK, Lakhani J, Benner R, Lele C, Patki K. A multicenter study of azithromycin, alone and in combination with chloroquine, for the treatment of acute uncomplicated Plasmodium falciparum malaria in India. J Infect Dis. 2005 May 15;191(10):1582-8. doi: 10.1086/429343. Epub 2005 Apr 11. PMID 15838784
- [Result] Mzayek F, Deng H, Mather FJ, Wasilevich EC, Liu H, Hadi CM, Chansolme DH, Murphy HA, Melek BH, Tenaglia AN, Mushatt DM, Dreisbach AW, Lertora JJ, Krogstad DJ. Randomized dose-ranging controlled trial of AQ-13, a candidate antimalarial, and chloroquine in healthy volunteers. PLoS Clin Trials. 2007 Jan 5;2(1):e6. doi: 10.1371/journal.pctr.0020006. PMID 17213921
- [Derived] Livezey J, Twomey P, Morrison M, Cicatelli S, Duncan EH, Hamer M, Lee C, Hutter J, Mills K, DeLuca J, Poon L, Selig D, Vuong C, Sousa J, Oliver T, Bennett J, Moon JE, Sikaffy A, Sedegah M, Tosh D, Kreishman-Deitrick M, Waterman P. An open label study of the safety and efficacy of a single dose of weekly chloroquine and azithromycin administered for malaria prophylaxis in healthy adults challenged with 7G8 chloroquine-resistant Plasmodium falciparum in a controlled human malaria infection model. Malar J. 2020 Sep 16;19(1):336. doi: 10.1186/s12936-020-03409-z. PMID 32938444